CLINICAL TRIAL: NCT01307046
Title: A Phase III, Randomized, Active-comparator Controlled Clinical Trial to Study the Efficacy and Safety of MK-0954A in Japanese Patients With Essential Hypertension Uncontrolled With the High Dose of Losartan Potassium
Brief Title: MK-0954A in Japanese Patients With Essential Hypertension Not Adequately Controlled With Losartan (MK-0954A-352)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0954A-352
Record Dates: First submitted 2011-03-01; First posted 2011-03-02 (Estimated); Results first posted 2013-03-22 (Estimated); Last update posted 2024-05-17 (Actual); Status verified 2022-02

CONDITIONS: Hypertension
Keywords: Essential hypertension; Uncontrolled hypertension; Antihypertensive agents; Blood pressure
MeSH Terms: conditions — Hypertension; Essential Hypertension | interventions — Losartan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- MK-0954A (Experimental): Participants administered MK-0954A, Placebo for Losartan 50 mg , and Placebo for Losartan 100 mg orally, once daily for 8 weeks.
  Interventions: Drug: MK-0954A; Drug: Placebo to losartan 100 mg; Drug: Placebo to losartan 50 mg
- Losartan (Active Comparator): Participants administered Losartan 100 mg, Placebo for MK-0954A, and Placebo for Losartan 50 mg orally, once daily for 8 weeks.
  Interventions: Drug: Losartan; Drug: Placebo to MK-0954A; Drug: Placebo to losartan 50 mg

INTERVENTIONS:
Drug: MK-0954A — Tablet containing losartan potassium (100 mg) and hydrochlorothiazide (12.5 mg), once daily
  Arms: MK-0954A
Drug: Losartan — Tablet containing losartan potassium (100 mg), once daily
  Arms: Losartan
Drug: Placebo to MK-0954A — Placebo tablet to match MK-0954A, once daily
  Arms: Losartan
Drug: Placebo to losartan 100 mg — Placebo tablet to match losartan 100 mg, once daily
  Arms: MK-0954A
Drug: Placebo to losartan 50 mg — Placebo tablet to match losartan 50 mg, once daily

SUMMARY:
This study is being conducted to evaluate the efficacy of MK-0954A in essential hypertension participants who are not adequately controlled with losartan.

ELIGIBILITY:
Inclusion criteria:

* Participant has a diagnosis of essential hypertension.
* Participant is not treated with antihypertensive medication and meets protocol-specified blood pressure criteria.
* Participant is treated with single antihypertensive medication, and meets protocol-specified blood pressure criteria.
* Participant is being treated with up to dual oral antihypertensive medications, and will be able to discontinue the prior antihypertensive medication.
* Participant has no clinically meaningful findings to be disqualified from the study at the discretion of the investigator.

Exclusion criteria:

* Regarding hypertension, participant is currently taking > 2 antihypertensive medications.
* Participant has a history of significant multiple and/or severe allergies to ingredients of Nu-lotan or Preminent and thiazide drug or related drug (i.e., sulfonamide-containing "chlortalidone" medicines)
* Participant is, at the time of signing informed consent, a user of recreational or illicit drugs or a recent history within the last year of drug or alcohol abuse or dependence.
* Participant is pregnant or breastfeeding or expecting to conceive or has a positive pregnancy test at the screening visit.
* Participant is currently participating or has participated in a study with an investigational compound (except losartan at any doses) or device within 30 days of signing informed consent.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 336 (Actual)
Dates: Start 2011-03-29 (Actual); Primary Completion 2012-02-07 (Actual); Study Completion 2012-02-07 (Actual)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Rakugi H, Tsuchihashi T, Shimada K, Numaguchi H, Nishida C, Yamaguchi H, Fujimoto G, Azuma K, Shirakawa M, Hanson ME, Fujita KP. Efficacy and safety of losartan 100 mg/hydrochlorothiazide 12.5 mg in Japanese subjects with essential hypertension: two randomized, controlled trials. Hypertens Res. 2014 Dec;37(12):1042-9. doi: 10.1038/hr.2014.114. Epub 2014 Jul 3. PMID 24990091

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | MK-0954A | Losartan
Started | 166 | 170
Completed | 154 | 159
Not Completed | 12 | 11
Not completed — Adverse Event | 3 | 3
Not completed — Lack of Efficacy | 0 | 2
Not completed — Physician Decision | 2 | 0
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Serum Potassium Withdrawal Criteria Met | 4 | 2
Not completed — Blood Pressure Withdrawal Criteria Met | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MK-0954A | Losartan | Total
Number analyzed (Participants) | 166 | 170 | 336
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.7 (9.2) | 54.9 (9.5) | 55.3 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 60 | 97
  Male | 129 | 110 | 239

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Trough Sitting Diastolic Blood Pressure (SiDBP)
Description: Sitting diastolic blood pressure was measured by automated sphygmomanometer pre-dose on Day 1 (baseline) and at 24 ± 2 hours after the last study drug administration (Day 56 ± 7 days).
Time Frame: Baseline and Week 8
Population: Full Analysis Set (FAS) population: defined as all randomized participants who received at least one dose of study treatment, had at least one post-randomization observation for the analysis endpoint subsequent
  to at least one dose of study treatment, and had baseline data for those analyses that required baseline data
Measure: Least Squares Mean (95% Confidence Interval); unit: mmHg
Arm/Group | MK-0954A | Losartan
Number analyzed (Participants) | 166 | 170
mmHg | -8.7 (0.6) [-9.9 to -7.6] | -3.6 (0.6) [-4.8 to -2.5]
Statistical Analysis 1: Comparison: MK-0954A vs Losartan; Test type: Superiority or Other; p < .001, constrained longitudinal data analysis; Difference in least square means = -5.1, 95% CI 2-sided [-6.8 to -3.4]

2. Secondary Outcome: Change From Baseline in Trough Sitting Systolic Blood Pressure (SiSBP)
Description: Sitting systolic blood pressure was measured by automated sphygmomanometer pre-dose on Day 1 (baseline) and at 24 ± 2 hours after the last study drug administration (Day 56 ± 7 days).
Time Frame: Baseline and Week 8
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mmHg
Arm/Group | MK-0954A | Losartan
Number analyzed (Participants) | 166 | 170
mmHg | -14.5 [-16.5 to -12.6] | -5.4 [-7.3 to -3.4]
Statistical Analysis 1: Comparison: MK-0954A vs Losartan; Test type: Superiority or Other; p < .001, constrained longitudinal data analysis; Difference in least square means = -9.2, 95% CI 2-sided [-11.9 to -6.5]

3. Primary Outcome: Percentage of Participants Who Experienced at Least One Adverse Event (AE)
Time Frame: 8 weeks
Population: All-Patients-as-Treated (APaT) Population: defined as all randomized participants who received at least one dose of study treatment.
Measure: Number; unit: percentage of participants
Arm/Group | MK-0954A | Losartan
Number analyzed (Participants) | 166 | 170
percentage of participants | 31.3 | 26.5

ADVERSE EVENTS:
Arm/Group | MK-0954A | Losartan
Serious Adverse Events (participants affected / at risk) | 0/166 | 0/170
Other Adverse Events (participants affected / at risk) | 9/166 | 9/170
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-0954A (N=166) | Losartan (N=170)
Nasopharyngitis (Infections and infestations) | 9 (11) | 9 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the sponsor as confidential must be deleted prior to submission. The sponsor review can be expedited to meet publication timelines.